CLINICAL TRIAL: NCT00196378
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Synthetic Conjugated Estrogens, B (Enjuvia) 0.3 mg Tablets for the Treatment of Vulvovaginal Atrophy in Healthy Postmenopausal Women
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Enjuvia 0.3 mg for the Treatment of Vulvovaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-ENJ-301
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2010-01

CONDITIONS: Menopause
Keywords: vaginal atrophy; vaginal dryness; vaginal itching; vaginal pain; dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — estrogens, conjugated synthetic B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Synthetic Conjugated estrogens, B
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Synthetic Conjugated estrogens, B — 1 (0.3mg) tablet daily
  Other Names: Enjuvia
  Arms: 1
Other: Placebo — 1 tablet daily
  Arms: 2

SUMMARY:
This is a two-arm, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy of Enjuvia 0.3 mg tablets for the treatment of moderate to severe symptoms of vulvovaginal atrophy in postmenopausal women with or without a hysterectomy and/or oophorectomy.

DETAILED DESCRIPTION:
The study will include a screening period up to 4 weeks and a 12-week treatment period. The overall study duration for participants will be approximately 16 weeks. Study participants will undergo physical and gynecological exams, and blood tests for clinical laboratory assessments. All patients with a uterus will undergo transvaginal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically postmenopausal
* Moderate or severe symptoms of vaginal atrophy (ie, dryness, itching, pain, uncomfortable intercourse)

Exclusion Criteria:

* Known sensitivity or contraindication to estrogens or progestins
* History or current diagnosis of endometrial hyperplasia
* Recent history of vaginal bleeding of unknown cause
* Recent history or diagnosis of endometriosis
* Any contraindication to estrogen therapy

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Mean change in the symptom identified by the patient to be most bothersome | Randomization to Week 12
Mean change in vaginal pH | Randomization to Week 12
Mean change in maturation index | Randomization to Week 12

SECONDARY OUTCOMES:
Safety and tolerability of Enjuvia | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Duraemd Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (34):
- United States (34):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Carmichael, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Gainesville, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Sarasota, Florida
  - Duramed Investigational Site, Venice, Florida
  - Duramed Investigational Site, Alpharetta, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Evansville, Indiana
  - Duramed Investigational Site, Baton Rouge, Louisiana
  - Duramed Investigational Site, Laurel, Maryland
  - Duramed Investigational Site, Billings, Montana
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Clarksville, Tennessee
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Fort Worth, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Sugarland, Texas
  - Duramed Investigational Site, Newport News, Virginia
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington

REFERENCES:
- [Derived] Simon JA, Reape KZ, Wininger S, Hait H. Randomized, multicenter, double-blind, placebo-controlled trial to evaluate the efficacy and safety of synthetic conjugated estrogens B for the treatment of vulvovaginal atrophy in healthy postmenopausal women. Fertil Steril. 2008 Oct;90(4):1132-8. doi: 10.1016/j.fertnstert.2007.07.1359. Epub 2007 Dec 3. PMID 18053998